CLINICAL TRIAL: NCT03166592
Title: Impact of Advanced Neuroimaging Techniques in Evaluation of Intra Axial Brain Masses Based on Magnetic Resonance Diagnostic Strategy in Adults
Brief Title: Evaluation of Intra Axial Brain Masses Based on Magnetic Resonance in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: IAM
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetic resonance imaging with contrast — injection of gadolinium contrast then acquisition of images with magnetic resonance imaging then spectroscopy

SUMMARY:
Although the Magnetic resonance imaging with contrast is the gold standard for diagnosis of intra axial brain masses. The conventional Magnetic resonance imaging appearances of intra axial brain masses can be non-specific and even the use of contrast agent is of limited benefit.

Contrast enhancement reflects only disruption of blood brain barrier. One third of high-grade malignancies are non-enhanced and may non-neoplastic lesions show contrast enhancement.

Reliable differentiation of neoplastic from non-neoplastic brain masses, or of high grade from low grade tumor, is difficult with conventional Magnetic resonance imaging

ELIGIBILITY:
1. Inclusion criteria:

   * An intra axial space occupying lesion/lesions detected on conventional structural imaging
2. Exclusion criteria:

   * MRI contraindications (as pace maker or claustrophobia).
   * Contrast hypersensitivity
   * Impaired renal function.
   * Pediatric age group

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All Magnetic resonance imaging detected brain cases referred from Neurosurgery & Neuropsychiatry departments as well as Outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with malignant masses | 1 hour
  sensitivity of the magnetic resonance spectroscopy in diagnosis of brain malignant masses

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Abbas, Assiut, Cairo Governorate
  - Assiut Faculty of Medicine, Asyut

IPD SHARING:
Plan to Share IPD: No